CLINICAL TRIAL: NCT02801591
Title: Effect of Recombinant Human Growth Hormone Injection on the Clinical Outcome of Poor Ovarian Response (POR) Clinical Outcome in Patients Undergoing in Vitro Fertilization / Embryo Transfer (IVF/ET)
Brief Title: Effect of Recombinant Human Growth Hormone Injection on the Clinical Outcome of POR in Patients Undergoing IVF/ET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Third Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GenSci GH AQ CT-POR
Record Dates: First submitted 2016-06-06; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Poor Ovarian Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GH AQ
  Interventions: Procedure: Conventional ovarian stimulation proctol without rhGH

INTERVENTIONS:
Procedure: Conventional ovarian stimulation proctol without rhGH

SUMMARY:
Observe the clinical efficacy and safety of Recombinant Human Growth Hormone Injection assisted in the treatment of the patients with poor ovarian response in vitro fertilization and embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 30-42 years old.
* Diagnosis of POR (2011 ESHRE Bologna Standard).
* At least two previous IVF failure history.
* Voluntarily to sign the "informed consent".

Exclusion Criteria:

* Severe acute and chronic liver and kidney disease，Such as liver cirrhosis, acute and chronic renal failure, hepatitis B virus activity period, etc.；Liver and kidney dysfunction.
* Endocrine and metabolic diseases，eg, diabetes、Thyroid function hyperthyroidism, Thyroid dysfunction, cushing's syndrome, hyperprolactinemia，hyperandrogenism.
* Related diseases affecting outcome of IVF pregnancy，eg, hydrosalpinx, hysteromyoma≥4cm, adenomyosis, stage III and IV endometriosis, untreated endometrial lesions, uterine malformation, genital tuberculosis, malignant tumor of reproductive system （include endometrial carcinoma, cervical carcinoma, ovarian cancer, fallopian tube carcinoma）.
* Allergic to E. coli expression product and its excipients.
* Subjects who participated in the past three months or are participating in other drug clinical researchers.
* IVF failure history≥3.
* The researchers consider who is not suitable for enrolling the group.

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Poor ovarian response
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | One year

SECONDARY OUTCOMES:
Number of retrieved oocytes | One year
Number of high quality embryos | One year
Number of embryos transferred | One year

CONTACTS AND LOCATIONS:
Overall Officials: Xin Na Chen, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing
  - People's Hospital of Peking University, Beijing